CLINICAL TRIAL: NCT04712136
Title: Healthy-related Quality of Life and Physical Activity of Children With Inherited Cardiac Arrhythmia or Inherited Cardiomyopathies: the Prospective Multicentre Controlled QUALIMYORYTHM Study
Brief Title: Healthy-related Quality of Life and Physical Activity of Children With Cardiac Malformations
Acronym: QUALIMYORYTHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Saint Pierre Institute - Palavas les Flots (Unknown); University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other); Hôpital Necker-Enfants Malades (Other); Hopital Lariboisière (Other); Nantes University Hospital (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL19-0554
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Long QT Syndrome; Brugada Syndrome; Catecholaminergic Polymorphic Ventricular Tachycardia; Arrhythmogenic Right Ventricular Dysplasia; Hypertrophic Cardiomyopathy; Dilated Cardiomyopathy; Restrictive Cardiomyopathy
Keywords: Life quality; Physical activity; Paediatric cardiology; Inherited cardiac arrhythmia; Genetic cardiomyopathies
MeSH Terms: conditions — Long QT Syndrome; Brugada Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Cardiomyopathy, Restrictive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac disease (Experimental): Children aged of 6 to 18 years old with an inherited cardiac arrhythmia (long QT syndrome, Brugada syndrome, catecholaminergic polymorphic ventricular tachycardia, or arrhythmogenic right ventricular dysplasia), or those with an inherited cardiomyopathy (hypertrophic, dilated, or restrictive cardiomyopathy).
  Interventions: Other: MRI
- Control group (Sham Comparator): Children aged 6 to 18 years old referred to the paediatric cardiology consultation who were classified in the control group after a completely normal check-up, including physical examination, electrocardiogram, and echocardiography.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI cardiac

SUMMARY:
The QUALIMYORYTHM trial is a multicentre controlled study, aiming to assess health-related quality of life (HRQoL) of 107 children aged 6 to 18 years old with inherited cardiac arrhythmia (long QT syndrome, Brugada syndrome, catecholaminergic polymorphic ventricular tachycardia, or arrhythmogenic right ventricular dysplasia), or inherited cardiomyopathies (hypertrophic, dilated, or restrictive cardiomyopathy), and to compare the results to those of 107 age and gender-matched healthy subjects. The secondary objective is to assess, in this population, the HRQoL according to disease characteristics, level of physical activity, exercise capacity, and socio-demographic data. Participants will wear a fitness tracker for 2 weeks.

DETAILED DESCRIPTION:
Advances in paediatric cardiology has improved the prognosis of children with inherited cardiac disorders. However, quality of life and physical activity have been scarcely analysed in children with inherited cardiac arrhythmia or inherited cardiomyopathies. Moreover, current guidelines on the eligibility of young athletes with inherited cardiac disorders for sports participation mainly rely on expert opinions and remain controversial.

The QUALIMYORYTHM trial is a multicentre controlled study. The main objective is to compare health-related quality of life (HRQoL) of children aged 6 to 18 years old with inherited cardiac arrhythmia (long QT syndrome, Brugada syndrome, catecholaminergic polymorphic ventricular tachycardia, or arrhythmogenic right ventricular dysplasia), or inherited cardiomyopathies (hypertrophic, dilated, or restrictive cardiomyopathy), to that of age and gender-matched healthy subjects. The secondary objective is to assess, in this population, HRQoL according to the disease clinical and genetic characteristics, the level of physical activity and motivation for sports, the exercise capacity (VO2max), and the socio-demographic data. Participants will wear a fitness tracker (actimeter watch) for 2 weeks. A total of 214 children are required to observe a significant difference of 7 ± 15 points in the PedsQL, with a power of 90% and an alpha risk of 5%.

The QUALIMYORYTHM trial intends to improve the level of evidence for future guidelines on sports eligibility in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 6 to 18 years old.
* Group 1: Patients with an inherited cardiac arrhythmia (long QT syndrome, Brugada syndrome, catecholaminergic polymorphic ventricular tachycardia, or arrhythmogenic right ventricular dysplasia), or those with an inherited cardiomyopathy (hypertrophic, dilated, or restrictive cardiomyopathy).
* Group 2: Children with a completely normal check-up, referred to the paediatric cardiology consultation for a non-severe functional symptom linked to exercise (murmur, palpitation, or dyspnoea) or for a medical sports certificate.
* Informed consent of parents or legal guardians, and oral assent of children

Exclusion Criteria:

* Patients who are not able to understand or fill out the questionnaires (QoL, physical activity and motivation questionnaires).
* Absolute contraindications for CPET: fever, uncontrolled asthma, respiratory failure, acute myocarditis or pericarditis, uncontrolled arrhythmias causing symptoms or haemodynamic compromise, uncontrolled heart failure, acute pulmonary embolus or pulmonary infarction, and children with mental impairment leading to inability to cooperate.
* Group 2: Children with any chronic disease, medical condition (cardiac, neurologic, respiratory, muscular, or renal), or medical treatment and those requiring any further specialized medical consultation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Total score of health-reported quality of life self questionnaire | baseline (1 day)
  PedsQL questionnaire

SECONDARY OUTCOMES:
The metabolic equivalent of task | during 14 days after inclusion
  measured by the wearable actimeter device.
physical activity level | baseline (1 day)
  Ricci and Gagnon questionnaire
Motivation towards health-oriented physical activity | baseline (1 day)
  EMAPS motivation scale
Exercise capacity | baseline (1 day)
  Cardiopulmonary exercise test with VO2max assessment
Myocardial morphologic assessment | baseline (1 day)
  cardiac MRI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Arnaud de Villeneuve, Montpellier, Occitanie, France

REFERENCES:
- [Background] Amedro P, Werner O, Abassi H, Boisson A, Souilla L, Guillaumont S, Calderon J, Requirand A, Vincenti M, Pommier V, Matecki S, De La Villeon G, Lavastre K, Lacampagne A, Picot MC, Beyler C, Delclaux C, Dulac Y, Guitarte A, Charron P, Denjoy-Urbain I, Probst V, Baruteau AE, Chevalier P, Di Filippo S, Thambo JB, Bonnet D, Pasquie JL. Health-related quality of life and physical activity in children with inherited cardiac arrhythmia or inherited cardiomyopathy: the prospective multicentre controlled QUALIMYORYTHM study rationale, design and methods. Health Qual Life Outcomes. 2021 Jul 28;19(1):187. doi: 10.1186/s12955-021-01825-6. PMID 34321045
- [Background] Souilla L, Avesani M, Boisson A, Requirand A, Matecki S, Vincenti M, Werner O, De La Villeon G, Pommier V, Pasquie JL, Guillaumont S, Amedro P. Cardiorespiratory fitness, muscle fitness, and physical activity in children with long QT syndrome: A prospective controlled study. Front Cardiovasc Med. 2023 Jan 11;9:1081106. doi: 10.3389/fcvm.2022.1081106. eCollection 2022. PMID 36712265
- [Background] Souilla L, Guillaumont S, Auer A, Metzler G, Requirand A, Vincenti M, De La Villeon G, Pasquie JL, Mottet D, Amedro P. Cardiac rehabilitation in children and adolescents with long QT syndrome: the RYTHMO'FIT pilot study. BMC Sports Sci Med Rehabil. 2024 Jul 12;16(1):152. doi: 10.1186/s13102-024-00941-2. PMID 38997778
- [Result] Souilla L, Werner O, Huguet H, Gavotto A, Vincenti M, Pasquie JL, De La Villeon G, Guillaumont S, Pommier V, Matecki S, Baruteau AE, Beyler C, Delclaux C, Denjoy I, Charron P, Chevalier P, Deliniere A, Andrianoely M, Cornuault L, Besnard-Neyraud C, Sacher F, Reant P, Mottet D, Picot MC, Amedro P; Quality of Life in Children With Inherited Cardiomyopathy or Arrhythmia (QUALIMYORYTHM) Study Group. Cardiopulmonary Fitness and Physical Activity Among Children and Adolescents With Inherited Cardiac Disease. JAMA Netw Open. 2025 Feb 3;8(2):e2461795. doi: 10.1001/jamanetworkopen.2024.61795. PMID 39998828